CLINICAL TRIAL: NCT00651638
Title: A Study of ARQ 197 in Healthy Volunteers to Assess the Pharmacokinetic (PK) Profile in Extensive and Poor Metabolizers as Defined by Cytochrome P450 2C19 (CYP 2C19) Genotype
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: ArQule, Inc., ArQule, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ARQ 197-112
Record Dates: First submitted 2008-03-27; First posted 2008-04-03 (Estimated); Last update posted 2008-06-19 (Estimated); Status verified 2008-06

CONDITIONS: Healthy
Keywords: PK and safety profile of ARQ 197
MeSH Terms: interventions — Therapeutics; ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Treatment with ARQ 197 — Treatment with ARQ 197

SUMMARY:
To assess the PK and safety profiles of ARQ 197 in extensive and poor metabolizers, as defined by CYP 2C19 genotype

DETAILED DESCRIPTION:
This is a pharmacokinetic study designed to compare the metabolism of ARQ 197 in normal healthy volunteers who are extensive metabolizers (EM) or poor metabolizers (PM) as defined by CYP 2C19 genotype. This is an open-label, single-dose, parallel group design in which healthy volunteer subjects will receive a single dose of ARQ 197

ELIGIBILITY:
Inclusion Criteria:

* Subject must provide written informed consent prior to any study related procedures
* Subjects must be between the ages of 18 and 65 years old
* Male participants must be surgically sterilized
* Female participants must be surgically sterilized or post menopausal and must have a negative serum pregnancy test. Post Menopausal is defined as at least one year without menses.
* Subject must, in the opinion of the Investigator, be willing and able to complete the study procedures

Exclusion Criteria:

* Subject must provide written informed consent prior to any study related procedures
* Subjects must be between the ages of 18 and 65 years old
* Male participants must be surgically sterilized
* Female participants must be surgically sterilized or post menopausal and must have a negative serum pregnancy test. Post Menopausal is defined as at least one year without menses.
* Subject must, in the opinion of the Investigator, be willing and able to complete the study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To assess the PK and safety profiles of ARQ 197 in extensive and poor metabolizers, as defined by CYP 2C19 genotype | May 2008

SECONDARY OUTCOMES:
To assess the effect of other CYP genotypes on the safety profile and PK profile of ARQ 197 | May 2008

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Kimberlin, MD, Principal Investigator — Covance Clinical Research Unit
Locations (1):
- Covance Clinical Research Unit, Inc., Evansville, Indiana, United States